CLINICAL TRIAL: NCT02272088
Title: Effect of Different Intensities of Exercise on Daily Energy Expenditure With Physical Activity in Overweight Boys
Acronym: PAPPAS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Rosely Sichieri, MD, PhD. Full Professor of Epidemiology, Rio de Janeiro State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IMS-NEBIN
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: physical activity; energy expenditure; compensatory mechanisms; adolescent
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- physical activity-moderate (Experimental): participants will be walking during 60 minutes in a moderate pace
  Interventions: Behavioral: physical activity-moderate; Behavioral: Intense physical activity
- intense physical activity (Experimental): participants will be running during 60 minutes in na intense pace.
  Interventions: Behavioral: physical activity-moderate; Behavioral: Intense physical activity

INTERVENTIONS:
Behavioral: physical activity-moderate — cross -over of moderate and intense physical activity
Behavioral: Intense physical activity — cross -over of moderate and intense physical activity

SUMMARY:
The main purpose of this study is evaluate the effect of different intensities of exercise (moderate vs. intense) on the daily energy expenditure in overweight adolescents.

DETAILED DESCRIPTION:
The specific objectives are:

1. Assess and quantify the existence of compensatory effect of exercise on subsequent physical activity.
2. Compare the amount of daily physical activity in adolescents subjected to different protocols of training intensity.

ELIGIBILITY:
Inclusion Criteria:

overweight 6th and 7th grades students consent form signed by parents / tutors

Exclusion Criteria:

diabetes mellitus hypertension or reported cardiovascular disease

Ages: 11 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
energy expenditure | one week
  measured by triaxial accelerometry

REFERENCES:
- [Derived] Paravidino VB, Mediano MFF, Sichieri R. Does a single bout of exercise influence subsequent physical activity and sedentary time in overweight boys? Physiol Behav. 2017 May 1;173:231-235. doi: 10.1016/j.physbeh.2017.02.016. Epub 2017 Feb 20. PMID 28223036
- [Derived] Paravidino VB, Mediano MF, Hoffman DJ, Sichieri R. Effect of Exercise Intensity on Spontaneous Physical Activity Energy Expenditure in Overweight Boys: A Crossover Study. PLoS One. 2016 Jan 15;11(1):e0147141. doi: 10.1371/journal.pone.0147141. eCollection 2016. PMID 26771742